CLINICAL TRIAL: NCT00522899
Title: The Effects of Mental Activity and Exercise on Cognitive Function in Older Adults Who Self-Report a Recent Decline in Memory or Thinking
Brief Title: The Mental Activity and eXercise Trial for Seniors
Acronym: MAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Alzheimer's Association (Other); National Institute on Aging (NIA) (NIH); Posit Science Corporation (Industry); YMCA of San Francisco (Unknown)
Responsible Party: Principal Investigator, Deborah Barnes, Associate Professor, Psychiatry and Epidemiology & Biostatistics, University of California, San Francisco
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: BarnesDeborahE-1; K01AG024069 (NIH); IIRG-06-27306 (Other Grant/Funding Number: Alzheimer's Association)
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Cognitive Impairment
Keywords: aged; exercise; cognitive therapy; dementia; prevention
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aerobic exercise (Experimental): Study-specific group exercise classes include 10' warm-up, 30' cardio, 5' cool down, 15' stretching/toning. Target heart rate is 60-75% of maximum. Study participants attend classes 60 min/day, 3 days/week for 12 weeks.
  Interventions: Behavioral: Group 1; Behavioral: Group 2
- Stretching/toning (Active Comparator): Study-specific stretching/toning exercise classes include 10' warm-up, 40' stretching/toning, 10' relaxation. Participants attend classes 60 minutes/day, 3 days/week for 12 weeks.
  Interventions: Behavioral: Group 3; Behavioral: Group 4
- Computer-based mental activity training (Experimental): Computer-based visual and auditory stimulation training programs developed by Posit Science corporation. Participants perform assigned mental activity on computers in their homes for 60 minutes/day, 3 days/week for 12 weeks.
  Interventions: Behavioral: Group 1; Behavioral: Group 3
- Educational DVD training (Active Comparator): Watching and listening to in-depth, college-level lectures on art, history and science on the computer. Participants perform assigned mental activities 60 minutes/day, 3 days/week for 12 weeks.
  Interventions: Behavioral: Group 2; Behavioral: Group 4

INTERVENTIONS:
Behavioral: Group 1 — Aerobic exercise plus computer-based mental activity training: both 3 days/week, 60 minutes/session for 12 weeks.
  Arms: Aerobic exercise; Computer-based mental activity training
Behavioral: Group 2 — Aerobic exercise plus educational DVDs: both 3 days/week, 60 minutes/session for 12 weeks.
  Arms: Aerobic exercise; Educational DVD training
Behavioral: Group 3 — Stretching/toning exercise group plus computer-based mental activity training: both 3 days/week, 60 minutes/session for 12 weeks.
  Arms: Computer-based mental activity training; Stretching/toning
Behavioral: Group 4 — Stretching/toning exercise group plus educational DVDs: both 3 days/week, 60 minutes/session for 12 weeks.
  Arms: Educational DVD training; Stretching/toning

SUMMARY:
The primary objective of this study is to conduct a randomized, controlled trial to determine whether engaging in mental activity or exercise, either alone or in combination, improves cognitive function in non-demented, inactive older adults who self-report a recent decline in memory or thinking. In addition, we, the researchers at the University of California, San Francisco, plan to seek funding to follow subjects over time to determine whether these interventions are associated with changes in rate of cognitive decline or risk of dementia after the intervention period has ended.

DETAILED DESCRIPTION:
SPECIFIC AIMS AND HYPOTHESES

Aim 1: To determine whether a 12-week, computer-based mental activity program improves cognitive function in non-demented, inactive elders.

We hypothesize that this mental activity program will improve cognitive function-especially visuospatial function-in non-demented, inactive elders.

Aim 2: To determine whether a 12-week exercise program improves cognitive function in non-demented, inactive elders.

We hypothesize that this exercise program will improve cognitive function-especially executive function-in non-demented, inactive elders.

Aim 3: To determine whether the effects of mental activity and exercise are additive or are more or less than the sum of their parts.

We hypothesize that the effects of these mental activity and exercise interventions will be additive.

Aim 4: To determine whether mental activity and/or exercise may slow cognitive decline or lower risk of dementia in non-demented, inactive elders.

We hypothesize that both mental activity and exercise will slow cognitive decline and lower risk of dementia, and that the effects will be greatest when mental activity and exercise are combined.

ELIGIBILITY:
Inclusion Criteria:

* Age > 64
* Self-report of recent decline in memory or thinking
* Low/no physical activity (<2 days/week for <30 minutes/session of moderate intensity activity over past 3 months)
* Low/no computer mental activity (<2 days/week for <30 minutes/session over past 3 months)
* Fluent in English
* Willingness to perform study activities

Exclusion Criteria:

* Evidence of dementia (based on self-report, physician diagnosis or score < 19 on Telephone Interview for Cognitive Status)
* Significant central nervous system disorder (Parkinson's disease, multiple sclerosis, ALS [Lou Gerig's disease])
* Major, current psychiatric disorder (major depressive disorder, schizophrenia, bipolar disorder, post-traumatic stress disorder, obsessive-compulsive disorder, psychiatric hospitalization in past 20 years)
* Major central nervous system event (stroke, transient ischemic attack/mini-stroke, seizure, or traumatic brain injury that has left a residual deficit)
* Significant heart disease (severe congestive heart failure, severe aortic stenosis, cardiac arrest, uncontrolled angina)
* Significant lung disease (requiring supplemental oxygen or oral or injected steroids)
* Other condition that would make participation potentially dangerous (cancer requiring treatment in past 3 years, severe arthritis, history of cardiac defibrillation, dialysis)
* Lack of physician approval
* Severe hearing or visual impairment
* History of learning disability
* Starting prescription medication to enhance cognitive function (e.g., memantine, aricept)
* Dependent in any basic activity of daily living (eating, dressing, bathing, toileting, getting out of bed/chair)
* History of alcohol abuse/heavy alcohol use
* History of drug abuse/heavy drug use
* Currently enrolled in another research study
* Fibromyalgia or tremor severe enough to prevent use of a computer mouse
* Planning to travel > 4 exercise class days during study period
* Behaviors during screening or baseline visit that, in the judgement of research staff, are likely to present significant problems (e.g., uncooperative, anger, inappropriate physical contact)
* Unable to perform neuropsychological evaluations
* Unable to complete consent process

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 126 (Actual)
Dates: Start 2007-08; Primary Completion 2009-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function summary score | 12 weeks

SECONDARY OUTCOMES:
Visual processing speed summary score (mental activity group), executive function summary score (exercise group), other measures (e.g., leisure activity, physical performance, physical function, depressive symptoms, sleep quality) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Barnes, PhD, MPH, Principal Investigator — University of California, San Francisco and San Francisco VA Medical Center
Locations (2):
- United States (2):
  - San Francisco Veterans Affairs Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

REFERENCES:
- [Derived] Barnes DE, Santos-Modesitt W, Poelke G, Kramer AF, Castro C, Middleton LE, Yaffe K. The Mental Activity and eXercise (MAX) trial: a randomized controlled trial to enhance cognitive function in older adults. JAMA Intern Med. 2013 May 13;173(9):797-804. doi: 10.1001/jamainternmed.2013.189. PMID 23545598